CLINICAL TRIAL: NCT03853278
Title: Developing and Testing a Self-management Support Intervention in Colorectal Cancer Survivors: A Mixed-methods Study
Brief Title: Self-management Support for Colorectal Cancer Survivors Colorectal Cancer Survivors: A Mixed-methods Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); Mackay Memorial Hospital (Other); Cathay General Hospital (Other)
Responsible Party: Principal Investigator, Tsae Jyy, Wang, RN PhD Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 107-2314-B-227-001-MY2
Record Dates: First submitted 2019-02-20; First posted 2019-02-25 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Neoplasms; self-management support; cancer survivor; healthy life styles
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The intervention includes a colorectal cancer self-management information booklet, a DVD, two individual skill training and 12 follow-up telephone calls. These are to establish participants' self-management skills and healthy lifestyle, including physical activity and healthy eating fruits and vegetables. The control group will receive health education leaflets.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization procedure was handled by an independent research assistant. Participants, care providers, investigator and outcomes assessors are blind to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- colorectal cancer self-management (Experimental): The intervention includes a colorectal cancer self-management information booklet, a DVD, two individual skill trainings and 12 follow-up telephone calls.These are to establish participants' self-management skills and healthy lifestyle, including physical activity and healthy eating fruits and vegetables.
  Interventions: Behavioral: colorectal cancer self-management
- No intervention control group (No Intervention): The control group will receive health education leaflets.

INTERVENTIONS:
Behavioral: colorectal cancer self-management — The intervention includes a colorectal cancer self-management information booklet, a DVD, two individual skill training and 12 follow-up telephone calls. These are to establish participants' self-management skills and healthy lifestyle, including physical activity and healthy eating fruits and vegetables.
  Arms: colorectal cancer self-management

SUMMARY:
Background: Survivors of colorectal cancer have to face long-term consequences of the disease and its treatment side effects, which in turn affect mood and psychological well-being. Self-management support may help colorectal cancer survivors to achieve healthy lifestyle and better adjustment.

However, there is little research evidence to support it and also no theory-based self-management support interventions specifically designed for colorectal cancer survivors in Taiwan.

Aim: The study aims is to test the efficacy of the Acceptance and Commitment Therapy -based self-management support program on the primary outcome, quality of life, and secondary outcomes, physical activity, fruit and vegetative intake, body mass index, sleep quality, emotion distress, and fatigue in colorectal cancer survivors .

Design: An experimental design with repeated measures will be used to test the intervention efficacy. A convenient sample of 250 colorectal cancer (stage I-III) survivors who has completed initial treatments will be recruited and randomized to the control or intervention group. The intervention includes a colorectal cancer self-management information booklet, a DVD, two individual skill trainings and 12 follow-up telephone calls. These are to establish participants' self-management skills and healthy lifestyle, including physical activity and healthy eating fruits and vegetables. The control group will receive health education leaflets. Outcome variables will be assessed on the baseline, 2th, 4th, and 6th month in both groups. Descriptive analysis will be used to describe patients' demographics, disease variables, and outcome variables. The Chi-square, t-test, and General Linear Mix-effect Model will be used to test the efficacy of the study interventions.

DETAILED DESCRIPTION:
Background: Colorectal cancer is the second most commonly diagnosed cancer in Taiwan. The five year relative survival rate of colorectal cancer is 61% and has become the third largest cancer survivor group. Survivors of colorectal cancer have to face long-term consequences of the disease and its treatment side effects, which in turn affect mood and psychological well-being. Overweight and unhealthy lifestyles will further impact on patient's prognosis and quality of life. The current follow-up systems often fail to adequately address patients' complex physical and mental needs. Self-management support may help colorectal cancer survivors to achieve healthy lifestyle and better adjustment. However, there is little research evidence to support it and also no theory-based self-management support interventions specifically designed for colorectal cancer survivors in Taiwan.

Aim: The study aims is to test the efficacy of the Acceptance and Commitment Therapy -based self-management support program on the primary outcome, quality of life, and secondary outcomes, physical activity, fruit and vegetative intake, body mass index, sleep quality, emotion distress, and fatigue in colorectal cancer survivors .

Design: An experimental design with repeated measures will be used to test the intervention efficacy. A convenient sample of 250 colorectal cancer (stage I-III) survivors who has completed initial treatments will be recruited and randomized to the control or intervention group. The intervention includes a colorectal cancer self-management information booklet, a DVD, two individual skill trainings and 12 follow-up telephone calls. These are to establish participants' self-management skills and healthy lifestyle, including physical activity and healthy eating fruits and vegetables. The control group will receive health education leaflets. Outcome variables will be assessed on the baseline, 2th, 4th, and 6th month in both groups.

Instruments: The study instruments include a body weight scale, Hospital Anxiety and Depression Scale, International Physical Activity Questionnaire, Eating at America's Table Study-Quick Food Scan, Pittsburgh Sleep Quality Index, FACIT-Fatigue, and FACT-C.

Data analysis: Descriptive analysis will be used to describe patients' demographics, disease variables, and outcome variables. The Chi-square, t-test, and General Linear Mix-effect Model will be used to test the efficacy of the study interventions.

Significance: The study results will provide evidence for the efficacy of the self-management support intervention for enhancing healthy life style and quality of life in colorectal cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnose with Colonrectal cancer (ICD-10 code: C18-C20, C21.8)
2. Stage I-III Colonrectal cancer
3. One month post curative cancer incision surgery for patients with cancer stage I-IIA
4. One month chemotherapy for patients with cancer stage IIB-III
5. Aged 20 and above
6. With the permission of the patient's doctor
7. Able to understand and sign the study inform consent

Exclusion Criteria:

1. The Eastern Cooperative Oncology Group ,( ECOG) performance score greater or equal to 3.
2. Diagnose with severe psychological diseases.
3. Life expectancy less than 3 month.
4. Had cancers before
5. Not able to communicate verbally or with writing

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy- Colorectal | Change from Baseline to 6 months
  There are two subscales, 27 items of FACT-General and 9 items of Colorectal Cancer Subscale. Each item is rated on a 5-point Likert scale (0-4). The total score of the 36 items represents the score of the scale. The possible score for the scale ranges from 0 to 136. The higher values represent better quality of life.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire | Change from Baseline to 6 months
  The Taiwan Version of International Physical Activity Questionnaire is used to measure a patient's physical activity. The scale has 7 items, asking patients the time they spent on walking, moderate, and vigorous physical activities during the past 7 days. The amounts of time spent on walking, moderate and vigorous physical activities are then multiplied by 3.3, 4.0, and 8.0 MET, respectively. The sum of the METs-min/wk for three types physically actives is the total score of the scale.
Eating at America's Table Study-Quick Food Scan | Change from Baseline to 6 months
  The scale measures a patient's intake of vegetables and fruits in the past month. There are 10 items in the scale, asking the amount and frequency of eating nine different types of vegetables and fruits. The frequency multiplied by the amount represents the total amount of vegetables and fruits consumed in the past month. The higher values indicate more vegetables and fruits patient consumed.
Body weight scale | Change from Baseline to 6 months
  The Body Mass Index (BMI) is calculated by the patient's body weight (kilograms) divided by height (meters) to the second power. Underweight is the BMI lower than18.5. Normal weight is the BMI higher or equal than18.5 and lower than 24. The overweight is the BMI higher or equal than 24 and lower than 27. The obese is the BMI higher or equal than 35.
Pittsburgh Sleep Quality Index | Change from Baseline to 6 months
  There are 10 items in the scale. Each item is rated on a 4-point Likert scale (0-3). The 10 items consist 7 dimensions. The total score of seven dimensions represents the scale score. The possible score for the scale ranges from 0 to 21. The higher values represent worse sleep quality.
Hospital Anxiety and Depression Scale | Change from Baseline to 6 months
  There are two subscales, HADS Anxiety and HADS Depression. Each subscale has 7 items. The possible score for each subscale scale ranges from 0 to 21. The higher values represent more anxiety or depression.
The Functional Assessment of Chronic Illness Therapy-Fatigue | Change from Baseline to 6 months
  There are 13 items in the scale. Each item is rated on a 5-point Likert scale (0-4). The total score of the 13 items represents the score of the scale. The possible score for the scale ranges from 0 to 52. The higher values represent more fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Tsae Jyy Wang, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (2):
- Taiwan (2):
  - Mackay Memorial Hospital, Taipei
  - Cathay General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aminisani N, Nikbakht H, Asghari Jafarabadi M, Shamshirgaran SM. Depression, anxiety, and health related quality of life among colorectal cancer survivors. J Gastrointest Oncol. 2017 Feb;8(1):81-88. doi: 10.21037/jgo.2017.01.12. PMID 28280612
- [Background] Siegel RL, Miller KD, Fedewa SA, Ahnen DJ, Meester RGS, Barzi A, Jemal A. Colorectal cancer statistics, 2017. CA Cancer J Clin. 2017 May 6;67(3):177-193. doi: 10.3322/caac.21395. Epub 2017 Mar 1. PMID 28248415
- [Background] Kim SH, Kim K, Mayer DK. Self-Management Intervention for Adult Cancer Survivors After Treatment: A Systematic Review and Meta-Analysis. Oncol Nurs Forum. 2017 Nov 1;44(6):719-728. doi: 10.1188/17.ONF.719-728. PMID 29052663
- [Derived] Wang TJ, Chang SC, Hsu HH, Huang CS, Lin TR, Lin YP, Chang KS. Efficacy of a self-management program on quality of life in colorectal cancer patients: A randomized controlled trial. Eur J Oncol Nurs. 2023 Dec;67:102431. doi: 10.1016/j.ejon.2023.102431. Epub 2023 Oct 30. PMID 37951069